CLINICAL TRIAL: NCT00058721
Title: SPECT Evaluation of Nicotinic Cholinergic Receptors in Parkinson's Disease
Brief Title: Single Photon Emission Computed Tomography to Study Receptors in Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030006; 03-N-0006
Record Dates: First submitted 2003-04-11; First posted 2003-04-11 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-01

CONDITIONS: Parkinson Disease
Keywords: Dementia; Feasibility; Dopamine; Lewy Body; Parkinson Disease; PD; Healthy Volunteer; HV
MeSH Terms: conditions — Parkinson Disease; Dementia

INTERVENTIONS:
Drug: I-123-5-IA85380

SUMMARY:
This study will use single photon emission computed tomography, or SPECT (see below), to examine brain nicotine receptors in evaluating the role of a chemical called acetylcholine in memory and other problems in Parkinson's disease (PD). Acetylcholine acts by binding to these nicotine receptors.

Healthy normal volunteers and patients with Parkinson's disease 40 years of age and older, with or without dementia, may be eligible for this study. Candidates will be screened with physical and neurological examinations, a pen and paper test of memory and other mental functions, blood tests, and, for women of childbearing potential, a pregnancy test. Patients with cognition problems will have more intensive mental function tests.

All participants will undergo the following procedures:

* Magnetic resonance imaging (MRI): This test uses a strong magnetic field and radio waves to show structural and chemical changes in the brain. During the scan, the subject lies on a table in a narrow cylinder (the scanner). The time required in the scanner is about 1 hour, during which the subject is asked to lie very still for 10 to 15 minutes at a time. He or she can speak with a staff member via an intercom system at all times during the procedure.
* SPECT: This nuclear medicine test produces a picture of the receptors in the brain. On the night before the scan, the day of the scan, and for 4 days after the scan, subjects take an oral dose of potassium iodide to protect the thyroid gland from the radioactive tracer used in the SPECT procedure. (People allergic to potassium iodide will take potassium perchlorate instead.) Before the scan, small radioactive markers containing 99Tc are glued to the subject's head. Two catheters (thin, flexible tubes) are placed in veins in the arms to inject the radioactive tracer [123I]5-I-A-85380 and to draw blood samples. Another catheter is placed in an artery in the wrist to draw arterial blood samples. During the scan, the subject lies on a bed with his or her head held still with a head holder. The scans are taken over a 6-hour period after injection of [123I]5-I-A-85380. An electrocardiogram, respiration, and blood pressure measures are taken before the tracer is injected, then 5 minutes after the injection, and again 30 to 60 minutes after the injection. Blood and urine samples are collected 5 to 6 hours after starting the scan. Participants are asked to urinate at least every 2 hours for 12 hours after injection of [123I]5-I-A-85380 to decrease radiation exposure.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is the second most common neurodegenerative disorder. PD is characterized primarily by motor impairment, but cognitive impairment is common and dementia may occur in up to 50% of patients. Cholinergic deficits have been widely demonstrated in PD patients with and without dementia. Cholinergic deficits are more profound in the setting of PD with dementia. The cholinergic system mediates aspects of learning and memory and deficits in cholinergic function are correlated with the degree of dementia in PD. Additionally, the cholinergic system may mediate certain aspects of motor function in PD. Data on cholinergic function, particularly relating to nicotinic cholinergic receptors, are limited to post mortem studies, and little is known about the role of the cholinergic system in vivo and how it relates to clinical phenomena. The aim of the current study is to assess the feasibility and usefulness of imaging of the high affinity alpha 4 beta 2 nicotinic cholinergic receptor in vivo, using SPECT (single photon emission computed tomography) imaging in patients with PD. The long-term goal of the present study is to further understanding of the role of the cholinergic system in the pathogenesis of PD and to elucidate potential diagnostic and therapeutic targets.

ELIGIBILITY:
INCLUSION CRITERIA -Patients:

Age greater than or equal to 40.

Diagnosis of PD.

Consent.

Responsible Caregiver (only for patients with dementia).

INCLUSION CRITERIA - Controls:

Age greater than or equal to 40.

Consent.

EXCLUSION CRITERIA - Patients and Controls:

Secondary cause of Parkinsonism, e.g. Wilson's disease, neuroleptic use.

Dementia not due to PD, abnormal screening labs for dementia

Or severe dementia with MMSE less than 15.

Neurological disorder other than PD that would effect protocol (e.g. stroke, Alzheimer's disease).

Use of cholinergic or anticholinergic agents within 60 days.

Abnormal MRI other than mild atrophy.

Claustrophobia.

Pregnancy or breast feeding.

Prior participation in other research protocols or clinical care in the last year such that radiation exposure would exceed the annual limits.

Any conditions that increase risk for MRI (pacemaker, metallic foreign body, etc.).

Any medical condition that in the opinion of the investigators would, interfere with the safe conduct of the study.

Both healthy subjects and patients will be excluded if they have more than moderate hypertension. The subject may be on anti-hypertensive medications. The initial screening must show no more than moderate hypertension- i.e. less than 160/95. On baseline evaluation on the day of the scan (i.e., before injection of tracer), the subject must be asymptomatic (no headache, dizziness, neurological symptoms, or blurred vision) AND have sustained BP less than 180/100.

History of smoking tobacco, use of nicotine gum or patch or other uses of nicotine within last 5 years.

Inability to provide consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 2003-04; Study Completion 2005-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Fujita M, Tamagnan G, Zoghbi SS, Al-Tikriti MS, Baldwin RM, Seibyl JP, Innis RB. Measurement of alpha4beta2 nicotinic acetylcholine receptors with [123I]5-I-A-85380 SPECT. J Nucl Med. 2000 Sep;41(9):1552-60. PMID 10994738
- [Background] Abreo MA, Lin NH, Garvey DS, Gunn DE, Hettinger AM, Wasicak JT, Pavlik PA, Martin YC, Donnelly-roberts DL, Anderson DJ, Sullivan JP, Williams M, Arneric SP, Holladay MW. Novel 3-Pyridyl ethers with subnanomolar affinity for central neuronal nicotinic acetylcholine receptors. J Med Chem. 1996 Feb 16;39(4):817-25. doi: 10.1021/jm9506884. PMID 8632405
- [Background] Charpantier E, Barneoud P, Moser P, Besnard F, Sgard F. Nicotinic acetylcholine subunit mRNA expression in dopaminergic neurons of the rat substantia nigra and ventral tegmental area. Neuroreport. 1998 Sep 14;9(13):3097-101. doi: 10.1097/00001756-199809140-00033. PMID 9804323